CLINICAL TRIAL: NCT04252547
Title: The Effect Of Kangaroo Mother Care On Test Weighing In Preterm Infants
Brief Title: Effect of Kangaroo Care on Test Weighing
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul University - Cerrahpasa (Other)
Responsible Party: Principal Investigator, Canan Genç, RN, Principal Investigator, Istanbul University - Cerrahpasa
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Supportive Care
Other Study IDs: 10840098-604.01.01-E.53511
Record Dates: First submitted 2020-01-09; First posted 2020-02-05 (Actual); Last update posted 2025-05-02 (Actual); Status verified 2025-01

CONDITIONS: Kangaroo Care; Weight Gain; Oxygen Saturation; Heart Rate
Keywords: kangaroo care; test weighing; Heart rate; oxygen saturation; preterm infants
MeSH Terms: conditions — Weight Gain | interventions — Kangaroo-Mother Care Method

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Grup 1 (Experimental): -"During the Procedure" Group 1 The preprocedural measurements(weight, heart rate and oxygen saturation ) will be applied to the infants in Group 1 before the first feeding hour when they are included in the study and then they will be held on their mothers' chest for skin-to-skin kangaroo care for half an hour. Their heart rate and oxygen saturation will be recorded for half an hour. At the end of the kangaroo care, the infant will be breastfed by his/her mother.
  During the second feeding hour, his/her heart rate and oxygen saturation will begin to be recorded ten minutes before the feeding hour. The data will be recorded for ten minutes and then the infant will be taken out of the incubator and weight is measured only in his/her clean diaper. He/she will be handed over to the mother to breastfeed.
  Interventions: Other: Kangaroo Care; Other: Control
- Grup 2 (Experimental): - "During the Procedure" Group 2 The preprocedural measurements will be applied to the infants in Group 2 before the first feeding hour when they are included in the study and then they will be breastfed by their mothers.
  The preprocedural measurements (weight, heart rate and oxygen saturation) will be applied to the infant during the second feeding hour and then he/she will be held on his/her mothers' chest for skin-to-skin kangaroo care for half an hour. Their heart rate and oxygen saturation will be recorded for half an hour. At the end of the kangaroo care, the infant will be breastfed by his/her mother.
  Interventions: Other: Kangaroo Care; Other: Control

INTERVENTIONS:
Other: Kangaroo Care — The preprocedural measurements (weight, heart rate, and oxygen saturation) will be recorded before the first feeding hour when they are included in the study and then they will be held on their mothers' chest for skin-to-skin kangaroo care for half an hour. Their heart rate and oxygen saturation will be recorded for half an hour. At the end of the kangaroo care, the infant will be breastfed by his/her mother. A chronometer will be started at that moment he/she begins sucking and terminated when he/she stops. The infant's heart rate and oxygen saturation will also continue to be recorded during the breastfeeding process. When the breastfeeding process is over, the infant will be allowed to rest in his/her mother's arms for two minutes and his/her physiological parameters will be recorded. Following the breastfeeding process, the infant will be weight is measured without a diaper change and his/her weight will be recorded. Then he/she will be taken back in the incubator to sleep.
Other: Control — The preprocedural measurements (weight, heart rate, and oxygen saturation) will be recorded before feeding when they are included in the study and then they will be breastfed by their mothers. The chronometer will be started at that moment he/she begins sucking and terminated when he/she stops. Also, the infant's heart rate and oxygen saturation will continue to be recorded during the breastfeeding process. When the breastfeeding process is over, the infant will be allowed to rest in his/her mother's arms for two minutes and his/her physiological parameters will be recorded. Following the breastfeeding process, the infant will be weighed without a diaper change and his/her weight will be recorded. When the care process is over, it will be taken back in the incubator to sleep.

SUMMARY:
The study will be conducted with the Crossover Randomized Controlled Method. The infants who have attained oral feeding in the neonatal intensive care unit will be divided into two groups via randomization in the computer environment. After the randomization, kangaroo care will be applied to the infants in Group 1 during the first feeding hour when they are included in the study and they will be breastfed by their mothers without any other application during the next feeding. On the other hand, no application will be performed on the infants in Group 2 during the first feeding hour when they are included in the study and kangaroo care will be applied to them during the second feeding hour. The infants in both groups will be breastfed by their mothers during the feeding hours.

DETAILED DESCRIPTION:
Test weighing is a feeding evaluation method which is used for evaluating the increase in infant's body weight and the amount of food intake before and after breastfeeding. Each gram is evaluated to be equivalent to one cc breast milk. The aim of the study is to evaluate the effect of kangaroo care applied to the preterm infants that have attained oral feeding and are breastfed by their mothers, on their physiological parameters, feeding condition and body weight increase. After weighing the infant only in his/her diaper before the feeding and applying kangaroo care in which skin-to-skin contact will be provided for half an hour, the mother will breastfeed the infant. The infant will be weighed once again after the feeding without diaper change and the effect of kangaroo care on test weighing and physiological parameters during the feeding process will be evaluated. Sample size of the study has been determined by the power analysis, in line with the results obtained from the studies which have been conducted using a similar research method. According to the analysis results, it has been calculated as 23 for each group and 46 in total. Parents of the infants meeting the study inclusion criteria will be informed both in written and verbally and then the study will be conducted with mothers who agree to participate in the study with their infants.

ELIGIBILITY:
Inclusion Criteria:

- Agreeing to participate in the study for parents.

The inclusion criteria for infants were as follows;

* Attaining to oral feeding by the physician in the neonatal intensive care unit
* Being born at 26-36+6 gestational week which is determined according to the mother's last period cycle
* Being at 32-39+6 postmenstrual week during the time they are included in the study
* Having body weight of 1500 grams and above
* Being breastfed at least once
* Having no health problems other than being preterm

Exclusion Criteria:

The exclusion criteria for infants were as follows;

* Suffering from gastrointestinal, neurological or genetic diseases (such as necrotizing enterocolitis, intracranial bleeding, hydrocephalia, omphalocele, down syndrome, gastroschisis) and other diseases
* Having a condition obstructing oral feeding (such as cleft palate, cleft lip, facial muscle paralysis, craniofacial abnormalities etc.)
* Receiving oxygen support

Ages: 32 Weeks to 40 Weeks | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 46 (Estimated)
Dates: Start 2024-06-09 (Actual); Primary Completion 2025-09-09 (Estimated); Study Completion 2026-01-09 (Estimated)

PRIMARY OUTCOMES:
Test Weighing | Change the body weight before feeding to after feeding at 1 day
  The infants' body weight before and after feeding will be measured using an 'Infant Scale'. The infants will be weighed naked only in their diaper before and after feeding, in order to evaluate the amount of milk they have received from their mothers' breast.

SECONDARY OUTCOMES:
Heart Rate | Change the Heart Rate 10 minutes before feeding to 2 minutes after feeding
  A device branded "Masimo Brand Radical 7 Pulse Oximetry" will be used to determine the infants' oxygen saturation and pulse rate. Heart rate of all the infants in Group 1 and Group 2 will begin to be recorded ten minutes before the first and second feeding hours when they are included in the study.
Oxygen Saturation | Change the Oxygen Saturation 10 minutes before feeding to 2 minutes after feeding
  A device branded "Masimo Brand Radical 7 Pulse Oximetry" will be used to determine the infants' oxygen saturation and pulse rate. Oxygen Saturation of all the infants in Group 1 and Group 2 will begin to be recorded ten minutes before the first and second feeding hours when they are included in the study.

CONTACTS AND LOCATIONS:
Overall Officials: Duygu Gözen, Assoc. Prof., Principal Investigator — Istanbul University Cerrahpaşa Florence Nightingale Faculty of Nursing; Ayhan Taştekin, prof., Principal Investigator — Istanbul Medipol University, Pediatrics
Locations (1):
- Istanbul Medipol University, Istanbul, Istanbul, Turkey (Türkiye)